CLINICAL TRIAL: NCT01592565
Title: An In-state Multi-center Evaluation of Treadmill Exercise Stress Cardiac Magnetic Resonance
Brief Title: Exercise Cardiac Magnetic Resonance Imaging Accuracy for Cardiovascular Stress Testing
Acronym: EXACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Karolina Zareba, MD, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007H0132 JD; NCT01504269 (obsolete NCT alias)
Record Dates: First submitted 2012-03-29; First posted 2012-05-07 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Diagnostic Cardiac Imaging — Cardiac Magnetic Resonance (CMR) offers superior image quality compared to echocardiography and nuclear imaging, and the ability to image both function and perfusion. Combining the superior image quality of CMR with the diagnostic information provided by exercise stress could result in a new, more accurate modality for diagnosing and evaluating coronary artery disease. This project is expected to show that CMR is at least equivalent to nuclear stress imaging and could potentially replace it in many instances, eliminating the need for radioisotope administration and the associated exposure of patients to ionizing radiation.

SUMMARY:
This study is being done to demonstrate a powerful new method for detecting heart disease that combines the proven prognostic capability of exercise stress testing with the superior image quality of Cardiac Magnetic Resonance Imaging (CMR). The investigators hope to demonstrate that exercise CMR has equivalent or superior diagnostic accuracy compared to exercise stress SPECT for detecting obstructive artery disease.

ELIGIBILITY:
Inclusion Criteria:

* any patient referred for stress SPECT
* known or suspected ischemic heart disease
* ability to perform adequate treadmill stress

Exclusion Criteria:

* any contraindication to MRI (e.g. ferromagnetic foreign body, cerebral aneurysm clip, pacemaker/ICD, severe claustrophobia)
* renal insufficiency (GFR < 40)
* known allergy to gadolinium-based contrast or iodinated contrast (because of the research CTA (computed tomography angiography) in patients not referred for cath after 2 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2010-08; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Exercise stress CMR has equivalent or superior diagnostic and prognostic value compared to exercise stress nuclear scintigraphy in patients suspected of CAD (coronary artery disease) | baseline
  Exercise nuclear and CMR examinations including aggregate assessment of exercise parameters, ECG findings, myocardial perfusion, segmental left ventricular wall motion (CMR only), and viability will be independently reviewed offline by a consensus of two reviewers blinded to the results of the other imaging study, and each test will be classified as either negative/adequate stress, negative/inadequate stress, positive for ischemia, or fixed abnormality/no ischemia.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Dickerson, MD, Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - The Lindner Center at The Christ Hospital, Cinncinatti, Ohio
  - The Ohio State University, Columbus, Ohio
  - University Of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Raman SV, Dickerson JA, Jekic M, Foster EL, Pennell ML, McCarthy B, Simonetti OP. Real-time cine and myocardial perfusion with treadmill exercise stress cardiovascular magnetic resonance in patients referred for stress SPECT. J Cardiovasc Magn Reson. 2010 Jul 12;12(1):41. doi: 10.1186/1532-429X-12-41. PMID 20624294
- [Background] Raman SV, Richards DR, Jekic M, Dickerson JA, Kander NH, Foster EL, Simonetti OP. Treadmill stress cardiac magnetic resonance imaging: first in vivo demonstration of exercise-induced apical ballooning. J Am Coll Cardiol. 2008 Dec 2;52(23):1884. doi: 10.1016/j.jacc.2008.08.046. No abstract available. PMID 19038687
- [Background] Foster EL, Arnold JW, Jekic M, Bender JA, Balasubramanian V, Thavendiranathan P, Dickerson JA, Raman SV, Simonetti OP. MR-compatible treadmill for exercise stress cardiac magnetic resonance imaging. Magn Reson Med. 2012 Mar;67(3):880-9. doi: 10.1002/mrm.23059. Epub 2011 Aug 16. PMID 22190228
- [Background] Jekic M, Foster EL, Ballinger MR, Raman SV, Simonetti OP. Cardiac function and myocardial perfusion immediately following maximal treadmill exercise inside the MRI room. J Cardiovasc Magn Reson. 2008 Jan 15;10(1):3. doi: 10.1186/1532-429X-10-3. PMID 18272005